CLINICAL TRIAL: NCT02066805
Title: Estimation of Off-Label Use of XGEVA® (Denosumab) Using Population-Based Databases in Denmark
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 20101335
Record Dates: First submitted 2014-02-13; First posted 2014-02-20 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: XGEVA Off-label Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: Database assessment of off-label XGEVA use

INTERVENTIONS:
Drug: Database assessment of off-label XGEVA use — No intervention is planned during this study as it involves analyses of patient electronic records from Northern Jutland Region and Copenhagen

SUMMARY:
This study aims to evaluate off-label XGEVA use in Denmark using data linked from registries and other sources in Northern Jutland Region and Copenhagen. This will allow for accurate assessment of prescriptions and diagnoses, especially those related to cancer patients during the first year post the initial market availability of XGEVA.

ELIGIBILITY:
Inclusion Criteria:

The study will include patients with a prescription for XGEVA® given in secondary care with a minimum of 108 XGEVA users, in the Northern Jutland Region and Copenhagen during the first 1-year post XGEVA market availability, defined as 12 months after RADS opinion on 24th January 2013 or after the minimum sample has been achieved.

Exclusion Criteria:

n/a

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include 108-200 patients who receive a prescription in secondary care of XGEVA during the first year after the initial market availability. These patients will be identified from the Danish National Registry of Patients and other sources in the Northern Jutland Region and Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
on or off label individual prescription type | 12 months
  Yes/no regarding whether an individual prescription was on (or off) label
on or off label patient treatment | 12 months
  Yes/no regarding whether the patient was treated on (or off) label

SECONDARY OUTCOMES:
type of off-label use | 12 months
  XGEVA prescription for each type of off-label use
off-label use stratified by administering department | 12 months
  Prescriptions that are for off-label use stratified by department that administers treatment

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com